CLINICAL TRIAL: NCT01077518
Title: Randomized Open Label of Ofatumumab and Bendamustine Combination Compared With Bendamustine Monotherapy in Indolent B-cell Non-Hodgkin's Lymphoma Unresponsive to Rituximab or a Rituximab-Containing Regimen During or Within Six Months of Treatment
Brief Title: Ofatumumab Bendamustine Combination Compared With Bendamustine Monotherapy in Indolent B-cell NHL Unresponsive to Rituxtherapy
Acronym: A+B
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated early as it did not meet the Primary efficacy objective after primary analysis.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110918; 2008-004177-17 (EudraCT Number); COMB157E2301 (Other: Novartis)
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Results first posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Lymphoma, Follicular
Keywords: Refractory; Safety; Efficacy; Rituximab refractory; Oncology; Ofatumumab; Bendamustine; Indolent B-cell Non- Hodgkin's Lymphoma Unresponsive; Rituximab; Rituximab-Containing Regimen
MeSH Terms: conditions — Lymphoma, Follicular; Neoplasms | interventions — ofatumumab

STUDY DESIGN:
Intervention Model Description: randomized open label bendamustine monotherapy vs. ofatumumab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ofatumumab and Bendamustine (Arm A) (Experimental): Up to 8 cycles of bendamustine (90 mg/m2) on Days 1,2 every 21 days with12 doses of ofatumumab (1000 mg, Day 1 q21 days when with bendamustine and q28 days when given as monotherapy)
  Interventions: Drug: Ofatumumab; Drug: Ofatumumab and Bendamustine infusions (Arm A)
- Bendamustine (Arm B) (Active Comparator): Up to 8 cycles of bendamustine (120 mg/m2) on Days 1,2 every 21 days
  Interventions: Drug: Ofatumumab; Drug: Bendamustine infusion; Drug: Bendamustine infusion (Arm B)

INTERVENTIONS:
Drug: Ofatumumab — Ofatumumab was a liquid concentrate solution for infusion presented in glass vials containing 50 mL of solution at a concentration of 20 mg/mL to provide 1000 mg per vial. The ofatumumab infusions were prepared in 1000 mL sterile, pyrogen-free 0.9% NaCl to yield a 1 mg/mL ofatumumab concentration infusion.
  Other Names: OMB157
Drug: Bendamustine infusion — Bendamustine 100 mg/vial, injection
  Arms: Bendamustine (Arm B)
Drug: Ofatumumab and Bendamustine infusions (Arm A) — Up to 8 cycles of Bendamustine (90 mg/m2 Days 1 and 2, every 21 days) given in combination with 12 doses of ofatumumab (1000 mg). Ofatumumab will be given on day 1 of each cycle of bendamustine as long as patients in Arm A receive bendamustine. Once patients in Arm A complete bendamustine therapy, the remaining doses of ofatumumab will be given monthly until all 12 doses are completed.
  Arms: Ofatumumab and Bendamustine (Arm A)
Drug: Bendamustine infusion (Arm B) — Bendamustine (120 mg/m2 Days 1 and 2, every 21 days, up to 8 cycles).
  Arms: Bendamustine (Arm B)

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of ofatumumab and bendamustine combination therapy in patients with indolent B-cell NHL that did not respond to rituximab or a rituximab-containing regimen during or within 6 months of the last rituximab treatment.

DETAILED DESCRIPTION:
Ofatumumab is an anti-CD20 monoclonal antibody shown to have monotherapy activity in patients with follicular lymphoma that has relapsed following rituximab-containing therapy. Bendamustine was approved by FDA for the treatment of in patients with indolent B-cell Non-Hodgkin's Lymphoma (NHL) that did not respond to rituximab or a rituximab-containing regimen during or within 6 months of the last rituximab treatment.

Biologics have demonstrated enhanced efficacy when added to chemotherapeutic combinations in the frontline treatment for indolent NHL. The combination of ofatumumab and bendamustine may provide additional clinical benefit and efficacy to those who no longer respond to rituximab or rituximab-containing regimens.

The objective of this study is to determine the effect of ofatumumab and bendamustine combination therapy in patients with indolent B-cell NHL that did not respond to rituximab or a rituximab-containing regimen during or within 6 months of the last rituximab treatment.

ELIGIBILITY:
Inclusion Criteria:

* Indolent lymphoma including Grades 1-3a follicular, small lymphocytic, lymphoplasmacytic, and marginal zone lymphoma; Stages III-IV, or bulky disease, Stage II. Tumor verified CD20+ and CT imaging done at screening verifying disease
* Indolent B-cell NHL that remains stable or unresponsive during or within 6 months of treatment with rituximab or a rituximab-containing regimen
* Indolent lymphoma including grades 1-3a follicular, small lymphocytic, lymphoplasmacytic, and marginal zone lymphoma; stages III-IV, or bulky disease stage II (i.e. as any single mass > 5 cm in any direction)
* ECOG Performance Status of 0, 1, or 2
* Life expectancy of at least 6 months
* 18 years or older
* Signed, written informed consent

Exclusion Criteria:

* Grade 3b follicular lymphoma or evidence that the indolent lymphoma has transformed to aggressive lymphoma
* Previous allogeneic stem cell transplant
* Previous autologous stem cell transplant, fludarabine therapy, or radioimmunotherapy in the past 12 months
* Previous external beam radiation therapy to the pelvis. Previous external beam radiation therapy for bony disease to the cranium, mediastinum, and axilla, or to two or to more than 3 vertebral bodies
* High dose steroids greater to or equal to 60 mg prednisone/day (or equivalent) within 3 months of randomization. No more than 10 mg prednisone (or equivalent) daily at the time of randomization
* Prior bendamustine treatment within 1 year of randomization not resulting in a CR or PR for at least 6 months
* Treatment with anti-CD20 monoclonal antibody within 3 months of randomization
* Known CNS involvement of indolent lymphoma
* Other past or current malignancy. Subjects free of malignancy for at least 5 years or have history of definitively treated non-melanoma skin cancer, or successfully treated in situ carcinoma, are eligible
* Chronic or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment
* Clinically significant cardiac disease
* History of significant cerebrovascular disease or event with significant symptoms
* Positive serology for Hepatitis B
* Current active liver or biliary disease (except Gibber's syndrome or asymptomatic gallstones, liver metastases, or otherwise stable chronic liver disease)
* Known HIV positive
* Abnormal/inadequate blood values, liver and kidney function
* Current participation in other clinical study
* Inability to comply with the protocol activities
* Lactating or pregnant women or female patients of child-bearing potential (or male patients with such partners) not willing to use adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2010-08-26 (Actual); Primary Completion 2018-01-03 (Actual); Study Completion 2018-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (130):
- United States (18):
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Palm Springs, California
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Coeur d'Alene, Idaho
  - Novartis Investigative Site, Silver Spring, Maryland
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Mineola, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Danville, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Morgantown, West Virginia
- Argentina (5):
  - Novartis Investigative Site, Capital Federal, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Derqui, Pilar, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
- Austria (7):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Leoben
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Steyr
  - Novartis Investigative Site, Vienna
- Belgium (4):
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Canada (5):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Barrie, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Saskatoon, Saskatchewan
- France (11):
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, La Roche-sur-Yon
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Saint-Denis
  - Novartis Investigative Site, Saint-Pierre
  - Novartis Investigative Site, Tours
- Germany (23):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Aschaffenburg, Bavaria
  - Novartis Investigative Site, Fürth, Bavaria
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Weilheim, Bavaria
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Giessen, Hesse
  - Novartis Investigative Site, Hanau, Hesse
  - Novartis Investigative Site, Kassel, Hesse
  - Novartis Investigative Site, Marburg, Hesse
  - Novartis Investigative Site, Bielefeld, North Rhine-Westphalia
  - Novartis Investigative Site, Bottrop, North Rhine-Westphalia
  - Novartis Investigative Site, Essen, North Rhine-Westphalia
  - Novartis Investigative Site, Goch, North Rhine-Westphalia
  - Novartis Investigative Site, Herford, North Rhine-Westphalia
  - Novartis Investigative Site, Leverkusen, North Rhine-Westphalia
  - Novartis Investigative Site, Paderborn, North Rhine-Westphalia
  - Novartis Investigative Site, Recklinghausen, North Rhine-Westphalia
  - Novartis Investigative Site, Kaiserslautern, Rhineland-Palatinate
  - Novartis Investigative Site, Koblenz, Rhineland-Palatinate
  - Novartis Investigative Site, Neunkirchen, Saarland
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bremen
- Greece (6):
  - Novartis Investigative Site, Alexandroupoli
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Haidari, Athens
  - Novartis Investigative Site, Heraklion, Crete
  - Novartis Investigative Site, Ioannina
  - Novartis Investigative Site, Piraeus
- Hong Kong (2):
  - Novartis Investigative Site, Shatin, New Territories
  - Novartis Investigative Site, Tuenmen
- Italy (10):
  - Novartis Investigative Site, San Giovanni Rotondo, Apulia
  - Novartis Investigative Site, Reggio Calabria, Calabria
  - Novartis Investigative Site, Napoli, Campania
  - Novartis Investigative Site, Meldola (FC), Emilia-Romagna
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Genoa, Liguria
  - Novartis Investigative Site, Milan, Lombardy
  - Novartis Investigative Site, Novara, Piedmont
  - Novartis Investigative Site, Terni, Umbria
  - Novartis Investigative Site, Verona, Veneto
- Japan (10):
  - Novartis Investigative Site, Aichi
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Hiroshima
  - Novartis Investigative Site, Hyōgo
  - Novartis Investigative Site, Ibaraki
  - Novartis Investigative Site, Kanagawa
  - Novartis Investigative Site, Miyagi
  - Novartis Investigative Site, Okayama
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Tokyo
- Poland (6):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Gdynia
  - Novartis Investigative Site, Legnica
  - Novartis Investigative Site, Opole
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Puerto Rico (2):
  - Novartis Investigative Site, Hato Rey
  - Novartis Investigative Site, San Juan
- Russia (12):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Kaluga
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Penza
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, St'Petersburg
  - Novartis Investigative Site, Tula
  - Novartis Investigative Site, Ufa
  - Novartis Investigative Site, Volgograd
- Novartis Investigative Site, Bratislava, Slovakia
- Ukraine (3):
  - Novartis Investigative Site, Kyiv
  - Novartis Investigative Site, Lviv
  - Novartis Investigative Site, Makiivka
- United Kingdom (5):
  - Novartis Investigative Site, Plymouth, Devon
  - Novartis Investigative Site, Northwood, Middlesex
  - Novartis Investigative Site, Harrow
  - Novartis Investigative Site, Southampton
  - Novartis Investigative Site, Uxbridge

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Rummel MJ, Janssens A, MacDonald D, Keating MM, Zaucha JM, Davis J, Lasher J, Babanrao Pisal C, Izquierdo M, Friedberg JW. A phase 3, randomized study of ofatumumab combined with bendamustine in rituximab-refractory iNHL (COMPLEMENT A + B study). Br J Haematol. 2021 Jun;193(6):1123-1133. doi: 10.1111/bjh.17420. Epub 2021 May 10. PMID 33973233

RESULTS

PARTICIPANT FLOW:
Groups:
- Ofa + Benda (Arm A): ofatumumab and bendamustine arm. Participants received up to 8 cycles of bendamustine (90 mg/m2) on Days 1,2 every 21 days with 12 doses of ofatumumab (1000 mg, Day 1 q21 days when with bendamustine and every 28 days
- Benda (Arm B): Bendamustine monotherapy. Participants received up to 8 cycles of bendamustine (120 mg/m2 on Days 1, 2 every 21 days
- Optional Ofa: Participants from the Benda arm who opted for optional ofatumumab therapy post disease progression.
Period: Treatment Phase - no Optional Ofa
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B) | Optional Ofa
Started | 173 | 173 | 0
Completed 5-year Follow-up | 64 | 64 | 0
Safety Population | 172 | 170 | 0
Completed | 95 | 108 | 0
Not Completed | 78 | 65 | 0
Not completed — Lost to Follow-up | 8 | 4 | 0
Not completed — Physician Decision | 10 | 11 | 0
Not completed — Study Terminated by Sponsor | 28 | 22 | 0
Not completed — Withdrawal by Subject | 32 | 28 | 0
Period: Optional Ofa Phase
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B) | Optional Ofa
Started | 0 | 0 | 32
Completed 5-year Follow-up | 0 | 0 | 12
Completed | 0 | 0 | 16
Not Completed | 0 | 0 | 16
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 12
Not completed — Withdrawal by Subject | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT):
Groups:
- Total: Total of all reporting groups
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B) | Total
Number analyzed (Participants) | 173 | 173 | 346
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (61.0) | 62.6 (63.0) | 62.2 (62.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 71 | 143
  Male | 101 | 102 | 203
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 6 | 16
  Not Hispanic or Latino | 163 | 167 | 330
  Unknown or Not Reported | 0 | 0 | 0
FLIPI-1 Score at Screening [Number; unit: participants] — Follicular Lymphoma International Prognostic Index-1 (FLIPI) is a prognostic tool that may be used to evaluate & select treatments based on differences in survival between risk groups. Low: (0 - 1) corresponds to better survival rate; intermediate: 2, corresponds to intermediate survival rate & high: (>=3) corresponds to worse survival rate. This index uses parameters related to subject characteristics such as age, tumor burden (Ann Arbor stage, number of nodal sites), tumor aggressiveness (serum Lactate Dehydrogenase (LDH) level), & consequences of the lymphoma on the host (hemoglobin level).
  participants
    0 - 2 | 100 | 93 | 193
    3 - 5 | 66 | 75 | 141
    Missing | 7 | 5 | 12
Baseline Absolute Lymphocyte Count (ALC) [Number; unit: Participants] — LLN - equal to the 5th percentile of a healthy, non-smoking population
  Participants
    < (Lower limit of normal (LLN) | 41 | 41 | 82
    >= LLN | 131 | 131 | 262
    Missing | 1 | 1 | 2
Fc Gamma Receptor (FcR) Gamma 3A Variation [Number; unit: Participants]
  GG | 21 | 18 | 39
  TG | 77 | 59 | 136
  TT | 61 | 62 | 123
  Missing | 14 | 34 | 48
Human Anti-Chimeric Antibodies (HACA) [Number; unit: Participants]
  Negative | 141 | 116 | 257
  Positive | 21 | 23 | 44
  Missing | 11 | 34 | 45

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) as Assessed by the Independent Review Committee (IRC)
Description: PFS is defined as the time interval between randomization until disease progression or death (due to any cause).
Time Frame: From randomization to the date of first documented disease progression or death due to any cause (67.5 months)
Population: ITT: The Intent-to-Treat (ITT) population included subjects who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 173 | 173
months | 16.66 [12.81 to 19.68] | 13.83 [11.30 to 16.89]
Statistical Analysis 1: Comparison: Ofa + Benda (Arm A) vs Benda (Arm B); Test type: Superiority; p = 0.1390, Stratified Log-Rank; Stratified Cox propor.hazards regression = 0.82, 95% CI 2-sided [0.62 to 1.07]

2. Secondary Outcome: Progression-free Survival (PFS) in Participants With Follicular Lymphoma (FL) Per IRC
Description: PFS is defined as the time interval between randomization until disease progression or death (due to any cause).
Time Frame: From randomization to the date of first documented disease progression or death due to any cause (67.5 months)
Population: Subjects in ITT with Follicular Lymphoma (FL). ITT population included subjects who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 120 | 119
months | 16.62 [11.17 to 20.47] | 12.12 [10.94 to 16.62]
Statistical Analysis 1: Comparison: Ofa + Benda (Arm A) vs Benda (Arm B); Test type: Other; p = 0.1076, Stratified Log-Rank; Stratified Cox propor.hazards regression = 0.76, 95% CI 2-sided [0.55 to 1.06]

3. Secondary Outcome: Overall Response Rate (ORR) in All Participants Per IRC
Description: ORR: Percentage of subjects achieving complete response (CR) or partial response (PR) from the start of randomization until disease progression or the start of new anti-cancer therapy, including the optional ofatumumab for subjects in Arm B based on responses from the IRC assessment of best overall response using the Revised Response Criteria for Malignant Lymphoma (RRCML). Response criteria is CR, PR, standard disease (SD), progressive disease (PD) or not estimable. CR is the complete disappearance of all detectable clinical evidence of disease & disease-related symptoms. PR is at least a 50% decrease from baseline in the sum of the product of the diameters (SPD) of target lesions. SD is failure to attain the criteria needed for a CR, PR or PD. PD is the appearance of any new lesion more than 1.5 cm in any axis or at least a 50% increase from nadir in the SPD of target or non target lesions or at least a 50% increase in the longest diameter(SLD) or any Target or non target lesions.
Time Frame: From randomization until the 217th PFS event occurred, up to about 67.5 months
Population: ITT: The ITT population included subjects who were randomized in the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 173 | 173
Percentage of participants | 73 [66 to 80] | 75 [67 to 81]
Statistical Analysis 1: Comparison: Ofa + Benda (Arm A) vs Benda (Arm B); for All participants; Test type: Other; p = 0.8003, Cochran-Mantel-Haenszel; adjusted for stratum

4. Secondary Outcome: Overall Response Rate (ORR) in Participants With FL Per IRC
Description: as for outcome 3
Time Frame: From randomization until the 217th PFS event occurred, up to about 67.5 months
Population: Subjects in ITT with FL. ITT population included subjects who were randomized in the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 120 | 119
Percentage of participants | 77 [68 to 84] | 76 [67 to 83]
Statistical Analysis 1: Comparison: Ofa + Benda (Arm A) vs Benda (Arm B); for Follicular Lymphoma (FL) participants; Test type: Other; p = 0.6130, Cochran-Mantel-Haenszel; adjusted for stratum

5. Secondary Outcome: Overall Survival (OS) in All Participants
Description: The interval of time between the date of randomization and the date of death due to any cause. For subjects who are alive, time of death will be censored at the date of last contact.
Time Frame: From randomization up to about 89 months
Population: ITT: The ITT population included subjects who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 173 | 173
months | 59.76 [46.63 to NA] — NA = Not evaluable because of a lot of censored data | 58.22 [36.44 to NA] — NA = Not evaluable because of a lot of censored data
Statistical Analysis 1: Comparison: Ofa + Benda (Arm A) vs Benda (Arm B); for All patients; Test type: Other; p = 0.4046, Stratified Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.62 to 1.21]

6. Secondary Outcome: Overall Survival (OS) in Participants With FL
Description: as for outcome 5
Time Frame: From randomization up to about 89 months
Population: Subjects in ITT with FL. ITT population included subjects who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 120 | 119
months | NA [45.60 to NA] — NA = Not evaluable because of a lot of censored data | 53.59 [36.44 to NA] — NA = Not evaluable because of a lot of censored data
Statistical Analysis 1: Comparison: Ofa + Benda (Arm A) vs Benda (Arm B); for FL participants; Test type: Superiority; p = 0.3768, Stratified Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.55 to 1.25]

7. Secondary Outcome: Time to Response in All Participants Per IRC
Description: Time to response = time from randomization to the first response (CR/ PR). If no CR/PR value was present data was to be censored at last adequate assessment.
Time Frame: From randomization to up to 67.5 months
Population: ITT: The ITT population included subjects who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 173 | 173
Months | 2.86 [2.83 to 2.92] | 2.89 [2.83 to 2.92]

8. Secondary Outcome: Time to Response in Participants With FL Per IRC
Description: as for outcome 7
Time Frame: From randomization to up to 67.5 months
Population: Subjects in ITT with FL. ITT population included subjects who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 120 | 119
Months | 2.86 [2.83 to 2.92] | 2.86 [2.83 to 2.89]

9. Secondary Outcome: Duration of Response in All Participants Per IRC
Description: Time (in months) from the initial response (CR/PR) to first documented sign of disease progression or death due to any cause.
Time Frame: time from the initial response (CR/PR) (Day 84) to first documented sign of disease progression or death due to any cause up to 67.5 months
Population: ITT: The ITT population included subjects who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 173 | 173
months | 17.71 [13.04 to 22.57] | 14.49 [10.84 to 16.76]

10. Secondary Outcome: Duration of Response in Participants With FL Per IRC
Description: as for outcome 9
Time Frame: as for outcome 9
Population: Subjects in ITT with FL. ITT population included subjects who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 120 | 119
months | 16.39 [11.53 to 20.53] | 11.20 [8.61 to 16.43]

11. Secondary Outcome: Time to Progression in All Participants Per IRC
Description: Time from randomization until disease progression
Time Frame: From randomization to the date of first documented disease progression, whichever occurred first, reported betwen day of first participant randomized up to about 67.5 months
Population: ITT: The ITT population included subjects who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 173 | 173
Months | 19.35 [14.32 to 23.10] | 16.56 [13.63 to 19.75]

12. Secondary Outcome: Time to Progression in Participants With FL Per IRC
Description: Time from randomization until disease progression
Time Frame: as for outcome 11
Population: Subjects in ITT with FL. ITT population included subjects who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 120 | 119
Months | 19.35 [14.16 to 24.87] | 13.80 [11.14 to 16.85]

13. Secondary Outcome: Time to Next Therapy in All Participants Per IRC
Description: Time to next therapy was defined as the time (in months) from randomization date to the date of receiving the next line treatment, including all therapy types.
Time Frame: from randomization date to the date of receiving the next line treatment or death, up to 67.5 months
Population: ITT: The ITT population included subjects who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 173 | 173
Months | 39.82 [28.81 to NA] — NA = Not evaluable because of a lot of censored data | 26.94 [21.72 to 39.75]

14. Secondary Outcome: Time to Next Therapy in Participants With FL Per IRC
Description: as for outcome 13
Time Frame: from randomization date to the date of receiving the next line treatment or death, up to 67.5 months
Population: Subjects in ITT with FL. ITT population included subjects who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 120 | 119
Months | 36.96 [23.79 to NA] — NA = Not evaluable because of a lot of censored data | 25.43 [18.37 to 47.70]

15. Secondary Outcome: PRO - Change From Baseline in Health Related Quality of Life (HRQL) Measures in All Participants: The FACT-Lym
Description: The Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) is intended as a lymphoma specific additional concerns subscale that is designed to supplement the FACT-G. The subscale consists of 15 items. Subjects respond to the items on a five point Likert scale ranging from 0 'Not at all' to 4 'Very much'. Subscale scores are calculated by summing individual items to obtain a score, then multiplying the sum of the item scores by the number of items in the subscale, then dividing by the number of items answered. The Score range is 0 -28 for Physical Well-Being, Social/Family Well-Being, 0 -24 for Functional Well-Being and 0 - 60 for the Lymphoma subscale (LYMS). FACT lymphoma TOI is the sum of Physical, Functional Well-Being & Lymphoma scores. FACT-G Total Score is the sum of Physical, Emotional, Social and Functional Well-Being scores. FACT-Lymph is the sum of Physical, Social, Emotional, Functional and Lymphoma scores. The higher the score, the better the QOL. C =cycle; D=Day
Time Frame: administered at the screening visit and C5D1 (month 5), C11D1 (month 11), D252, 12m post-D252, withdrawal (24m post-D252) up to 67.5 months; Cycle = 21 days
Population: ITT: The ITT population included subjects who were randomized in the study.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 173 | 173
scores on a scale
  Physical well-being score: C5D1: number analyzed (Participants) | 126 | 118
  Physical well-being score: C5D1 | 0.2 (4.36) | -2.8 (5.54)
  Physical well-being score C11D1: number analyzed (Participants) | 104 | 78
  Physical well-being score C11D1 | 1.1 (4.58) | 1.0 (4.25)
  Physical well-being score D252: number analyzed (Participants) | 3 | 6
  Physical well-being score D252 | -5.0 (9.64) | 1.7 (9.18)
  Physical well-being score 12M post-D252: number analyzed (Participants) | 67 | 53
  Physical well-being score 12M post-D252 | 0.9 (5.59) | 1.3 (4.52)
  Physical well-being score Withdrawal: number analyzed (Participants) | 12 | 15
  Physical well-being score Withdrawal | -4.1 (6.78) | -1.5 (6.61)
  Social/Family well-being score C5D1: number analyzed (Participants) | 126 | 118
  Social/Family well-being score C5D1 | 0.2 (4.94) | -0.5 (5.24)
  Social/Family well-being score C11D1: number analyzed (Participants) | 104 | 78
  Social/Family well-being score C11D1 | -1.2 (6.09) | -1.1 (6.45)
  Social/Family well-being score D252: number analyzed (Participants) | 3 | 6
  Social/Family well-being score D252 | -1.6 (3.24) | -5.4 (9.08)
  Soc./Fam. well-being score 12M post-D252: number analyzed (Participants) | 67 | 53
  Soc./Fam. well-being score 12M post-D252 | 0.3 (5.21) | -1.3 (4.81)
  Social/Family well-being score Withdrawal: number analyzed (Participants) | 12 | 15
  Social/Family well-being score Withdrawal | 0.9 (7.69) | 0.3 (3.53)
  Emotional well-being score C5D1: number analyzed (Participants) | 126 | 118
  Emotional well-being score C5D1 | 1.7 (3.97) | 0.1 (4.10)
  Emotional well-being score C11D1: number analyzed (Participants) | 103 | 78
  Emotional well-being score C11D1 | 1.4 (4.12) | 0.7 (3.90)
  Emotional well-being score D252: number analyzed (Participants) | 3 | 6
  Emotional well-being score D252 | -5.3 (2.08) | -2.5 (5.89)
  Emotional well-being score 12M post-D252: number analyzed (Participants) | 67 | 53
  Emotional well-being score 12M post-D252 | 1.5 (4.45) | 0.7 (4.15)
  Emotional well-being score Withdrawal: number analyzed (Participants) | 12 | 15
  Emotional well-being score Withdrawal | -2.2 (4.80) | -2.3 (4.12)
  Functional well-being score C5D1: number analyzed (Participants) | 126 | 118
  Functional well-being score C5D1 | 0.7 (5.08) | -1.5 (5.79)
  Functional well-being score C11D1: number analyzed (Participants) | 103 | 78
  Functional well-being score C11D1 | 1.1 (5.62) | -0.6 (5.52)
  Functional well-being score D252: number analyzed (Participants) | 3 | 6
  Functional well-being score D252 | -4.3 (5.69) | -2.2 (13.76)
  Functional well-being score 12M post-D252: number analyzed (Participants) | 67 | 53
  Functional well-being score 12M post-D252 | 1.1 (4.82) | 0.8 (5.55)
  Functional well-being score Withdrawal: number analyzed (Participants) | 12 | 15
  Functional well-being score Withdrawal | -2.3 (4.27) | -1.6 (6.47)
  Lymphoma subscale score C5D1: number analyzed (Participants) | 126 | 118
  Lymphoma subscale score C5D1 | 3.6 (7.88) | -1.0 (9.65)
  Lymphoma subscale score C11D1: number analyzed (Participants) | 104 | 78
  Lymphoma subscale score C11D1 | 4.4 (8.88) | 2.3 (6.53)
  Lymphoma subscale score D252: number analyzed (Participants) | 3 | 6
  Lymphoma subscale score D252 | -2.3 (14.98) | 0.7 (18.22)
  Lymphoma subscale score 12M post-D252: number analyzed (Participants) | 67 | 53
  Lymphoma subscale score 12M post-D252 | 3.2 (7.77) | 2.0 (7.71)
  Lymphoma subscale score Withdrawal: number analyzed (Participants) | 12 | 15
  Lymphoma subscale score Withdrawal | -1.4 (6.16) | -1.6 (7.65)
  FACT-Lymphoma TOI C1D1: number analyzed (Participants) | 126 | 118
  FACT-Lymphoma TOI C1D1 | 4.5 (14.64) | -5.3 (18.67)
  FACT-Lymphoma TOI C11D1: number analyzed (Participants) | 103 | 78
  FACT-Lymphoma TOI C11D1 | 6.7 (15.84) | 2.7 (13.24)
  FACT-Lymphoma TOI D252: number analyzed (Participants) | 3 | 6
  FACT-Lymphoma TOI D252 | -11.7 (28.75) | 0.2 (36.56)
  FACT-Lymphoma TOI 12M post-D252: number analyzed (Participants) | 67 | 53
  FACT-Lymphoma TOI 12M post-D252 | 5.1 (15.94) | 4.1 (14.62)
  FACT-Lymphoma TOI Withdrawal: number analyzed (Participants) | 12 | 14
  FACT-Lymphoma TOI Withdrawal | -7.8 (14.55) | -4.3 (16.77)
  FACT-G Total Score C5D1: number analyzed (Participants) | 126 | 118
  FACT-G Total Score C5D1 | 2.7 (12.82) | -4.7 (15.26)
  FACT-G Total Score C11D1: number analyzed (Participants) | 103 | 78
  FACT-G Total Score C11D1 | 2.3 (13.00) | 0.1 (14.11)
  FACT-G Total score D252: number analyzed (Participants) | 3 | 6
  FACT-G Total score D252 | -16.2 (15.71) | -8.4 (31.22)
  FACT-G Total Score 12M post-D252: number analyzed (Participants) | 67 | 53
  FACT-G Total Score 12M post-D252 | 3.7 (13.75) | 1.5 (13.44)
  FACT-G Total Score Withdrawal: number analyzed (Participants) | 12 | 15
  FACT-G Total Score Withdrawal | -7.7 (11.91) | -5.3 (13.10)
  FACT-Lymph. Tot. score C5D1: number analyzed (Participants) | 126 | 118
  FACT-Lymph. Tot. score C5D1 | 6.3 (18.78) | -5.8 (23.05)
  FACT-Lymph. Tot. score C11D1: number analyzed (Participants) | 103 | 78
  FACT-Lymph. Tot. score C11D1 | 6.7 (18.95) | 2.4 (18.73)
  FACT-Lymph. Tot. score D252: number analyzed (Participants) | 3 | 6
  FACT-Lymph. Tot. score D252 | -18.6 (30.50) | -7.7 (44.64)
  FACT-Lymph. Tot. score 12M post-D252: number analyzed (Participants) | 67 | 53
  FACT-Lymph. Tot. score 12M post-D252 | 6.9 (19.78) | 3.5 (18.77)
  FACT-Lymph. Tot. score Withdrawal: number analyzed (Participants) | 12 | 14
  FACT-Lymph. Tot. score Withdrawal | -9.1 (15.96) | -6.5 (18.53)

16. Secondary Outcome: PRO - Change From Baseline in Health Related Quality of Life (HRQL) Measures in Participants With FL: The FACT-Lym
Description: as for outcome 15
Time Frame: administered at the screeing visit and C5D1 (month 5), C11D1 (month 11), D252, 12m post-D252, withdrawal (24m post-D252) up to 67.5 months; Cycle = 21 days
Population: Subjects in ITT with FL. ITT population included subjects who were randomized in the study.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 120 | 119
scores on a scale
  Physical well-being score C5D1: number analyzed (Participants) | 87 | 78
  Physical well-being score C5D1 | 0.0 (4.66) | -3.4 (5.87)
  Physical well-being score C11D1: number analyzed (Participants) | 72 | 47
  Physical well-being score C11D1 | 0.9 (4.16) | 1.2 (4.74)
  Physical well-being score D252: number analyzed (Participants) | 1 | 2
  Physical well-being score D252 | 2.0 (NA) — NA = Standard Deviation not available since only 1 participant was analyzed for the assessment | 7.5 (17.68)
  Physical well-being score 12M post-D252: number analyzed (Participants) | 48 | 30
  Physical well-being score 12M post-D252 | 0.5 (6.15) | 1.8 (4.37)
  Physical well-being score Withdrawal: number analyzed (Participants) | 6 | 11
  Physical well-being score Withdrawal | -5.0 (7.64) | -0.6 (6.31)
  Social/Family well-being score C5D1: number analyzed (Participants) | 87 | 78
  Social/Family well-being score C5D1 | -0.1 (4.38) | -0.7 (5.48)
  Social/Family well-being score C11D1: number analyzed (Participants) | 72 | 47
  Social/Family well-being score C11D1 | -1.6 (5.38) | -1.4 (5.61)
  Social/Family well-being score D252: number analyzed (Participants) | 1 | 2
  Social/Family well-being score D252 | 2.0 (NA) — NA = Standard Deviation not available since only 1 participant was analyzed for the assessment | 2.5 (3.54)
  Soc./Fam. well-being score 12M post-D252: number analyzed (Participants) | 48 | 30
  Soc./Fam. well-being score 12M post-D252 | 0.3 (5.35) | -1.9 (5.14)
  Social/Family well-being score Withdrawal: number analyzed (Participants) | 6 | 11
  Social/Family well-being score Withdrawal | 1.1 (5.79) | 0.6 (2.57)
  Emotional well-being score C5D1: number analyzed (Participants) | 87 | 78
  Emotional well-being score C5D1 | 1.8 (3.65) | -0.0 (4.41)
  Emotional well-being score C11D1: number analyzed (Participants) | 72 | 47
  Emotional well-being score C11D1 | 1.2 (4.30) | 0.5 (4.10)
  Emotional well-being score D252: number analyzed (Participants) | 1 | 2
  Emotional well-being score D252 | -6.0 (NA) — NA = Standard Deviation not available since only 1 participant was analyzed for the assessment | -1.0 (9.90)
  Emotional well-being score 12M post-D252: number analyzed (Participants) | 48 | 30
  Emotional well-being score 12M post-D252 | 1.5 (4.85) | 0.6 (2.68)
  Emotional well-being score Withdrawal: number analyzed (Participants) | 6 | 11
  Emotional well-being score Withdrawal | -2.3 (5.28) | -1.9 (4.59)
  Functional well-being score C5D1: number analyzed (Participants) | 87 | 78
  Functional well-being score C5D1 | 0.1 (4.58) | -1.7 (5.74)
  Functional well-being score C11D1: number analyzed (Participants) | 72 | 47
  Functional well-being score C11D1 | 0.5 (4.99) | -0.0 (4.84)
  Functional well-being score D252: number analyzed (Participants) | 1 | 2
  Functional well-being score D252 | -6.0 (NA) — NA = Standard Deviation not available since only 1 participant was analyzed for the assessment | 7.0 (15.56)
  Functional well-being score 12M post-D252: number analyzed (Participants) | 48 | 30
  Functional well-being score 12M post-D252 | 0.7 (4.99) | 1.0 (5.75)
  Functional well-being score Withdrawal: number analyzed (Participants) | 6 | 11
  Functional well-being score Withdrawal | -1.6 (4.06) | -1.5 (7.15)
  Lymphoma subscale score C5D1: number analyzed (Participants) | 87 | 78
  Lymphoma subscale score C5D1 | 3.7 (7.33) | -2.2 (9.71)
  Lymphoma subscale score C11D1: number analyzed (Participants) | 72 | 47
  Lymphoma subscale score C11D1 | 3.7 (8.70) | 2.4 (6.79)
  Lymphoma subscale score D252: number analyzed (Participants) | 1 | 2
  Lymphoma subscale score D252 | -18.7 (NA) — NA = Standard Deviation not available since only 1 participant was analyzed for the assessment | 7.0 (38.18)
  Lymphoma subscale score 12M post-D252: number analyzed (Participants) | 48 | 30
  Lymphoma subscale score 12M post-D252 | 2.6 (8.00) | 2.2 (6.63)
  Lymphoma subscale score Withdrawal: number analyzed (Participants) | 6 | 11
  Lymphoma subscale score Withdrawal | -2.5 (6.76) | -0.4 (7.17)
  FACT-Lymphoma TOI C5D1: number analyzed (Participants) | 87 | 78
  FACT-Lymphoma TOI C5D1 | 3.7 (13.51) | -7.3 (18.77)
  FACT-Lymphoma TOI C11D1: number analyzed (Participants) | 72 | 47
  FACT-Lymphoma TOI C11D1 | 5.0 (14.74) | 3.6 (14.01)
  FACT-Lymphoma TOI D252: number analyzed (Participants) | 1 | 2
  FACT-Lymphoma TOI D252 | -2.0 (NA) — NA = Standard Deviation not available since only 1 participant was analyzed for the assessment | 21.5 (71.42)
  FACT-Lymphoma TOI 12M post-D252: number analyzed (Participants) | 48 | 30
  FACT-Lymphoma TOI 12M post-D252 | 3.7 (16.94) | 4.9 (12.32)
  FACT-Lymphoma TOI Withdrawal: number analyzed (Participants) | 6 | 10
  FACT-Lymphoma TOI Withdrawal | -9.2 (15.40) | -1.7 (15.26)
  FACT-G Total score C5D1: number analyzed (Participants) | 87 | 78
  FACT-G Total score C5D1 | 1.7 (11.40) | -5.8 (16.32)
  FACT-G Total score C11D1: number analyzed (Participants) | 72 | 47
  FACT-G Total score C11D1 | 1.0 (12.17) | 0.2 (13.96)
  FACT-G Total score D252: number analyzed (Participants) | 1 | 2
  FACT-G Total score D252 | -8.0 (NA) — NA = Standard Deviation not available since only 1 participant was analyzed for the assessment | 16.0 (39.60)
  FACT-G Total score 12M post-D252: number analyzed (Participants) | 48 | 30
  FACT-G Total score 12M post-D252 | 2.9 (14.62) | 1.4 (11.25)
  FACT-Lymphoma Tot. score C5D1: number analyzed (Participants) | 87 | 78
  FACT-Lymphoma Tot. score C5D1 | 5.4 (16.55) | -8.0 (24.11)
  FACT-Lymphoma Tot. score C11D1: number analyzed (Participants) | 72 | 47
  FACT-Lymphoma Tot. score C11D1 | 4.7 (17.52) | 2.7 (19.60)
  FACT-Lymphoma Tot. score D252: number analyzed (Participants) | 1 | 2
  FACT-Lymphoma Tot. score D252 | -6.0 (NA) — NA = Standard Deviation not available since only 1 participant was analyzed for the assessment | 23.0 (77.78)
  FACT-Lymphoma Tot. score 12M post-D252: number analyzed (Participants) | 48 | 30
  FACT-Lymphoma Tot. score 12M post-D252 | 5.5 (20.73) | 3.6 (14.44)
  FACT-Lymphoma Tot. score Withdrawal: number analyzed (Participants) | 6 | 10
  FACT-Lymphoma Tot. score Withdrawal | -10.4 (15.02) | -3.1 (18.48)

17. Secondary Outcome: PRO - Change From Baseline in HRQL Measures in All Participants: The EQ-5D
Description: The EuroQoL Five-Dimension (EQ-5D) is a self-administered, generic, indirect utility measure used for health economic analysis.EQ-5D should be answered as one of 3 levels about current condition for 5 dimensions and was calculated total average by giving a weighting on 3 level of answers (EQ-5D levels into 'no problems' (level 1) and 'problems' (level 2 and 3)).
  Table of scores by each level for EQ-5D items: mobility(level 1=0, level2=0.069,level 3=0.314), self care(level 1=0, level2=0.104,level 3=0.214), usual activities(level 1=0, level2=0.036,level 3=0.094), pain/discomfort (level 1=0, level2=0.,level 3=0.386) and anxiety/depression(level 1=0, level2=0.071,level 3=0.2)
  *EQ-5D Total = 1 - 0.081 - (the score of the each level) - 0.269 (if at least one of level 3 presents)
Time Frame: administered at screening and C5D1 (month 5), C11D1 (month 11), D252, 12m post-D252, withdrawal (24m post-D252) up to 67.5 months; Cycle = 21 days
Population: ITT: The ITT population included subjects who were randomized in the study.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 173 | 173
scores on a scale
  EQ5D01-EQ VAS Score C5D1: number analyzed (Participants) | 124 | 115
  EQ5D01-EQ VAS Score C5D1 | 5.8 (18.10) | -3.8 (19.25)
  EQ5D01-EQ VAS Score C11D1: number analyzed (Participants) | 101 | 78
  EQ5D01-EQ VAS Score C11D1 | 12.9 (19.38) | 2.7 (18.96)
  EQ5D01-EQ VAS Score D252: number analyzed (Participants) | 3 | 6
  EQ5D01-EQ VAS Score D252 | -11.7 (16.07) | -0.8 (19.66)
  EQ5D01-EQ VAS Score 12M post-D252: number analyzed (Participants) | 65 | 52
  EQ5D01-EQ VAS Score 12M post-D252 | 14.7 (19.71) | 7.1 (19.14)
  EQ5D01-EQ VAS Score Withdrawal: number analyzed (Participants) | 12 | 15
  EQ5D01-EQ VAS Score Withdrawal | -14.7 (17.03) | 0.7 (34.41)
  EuroQoL Tariffs C5D1: number analyzed (Participants) | 122 | 116
  EuroQoL Tariffs C5D1 | 0.21 (0.24) | 0.0 (0.22)
  EuroQoL Tariffs C11D1: number analyzed (Participants) | 102 | 78
  EuroQoL Tariffs C11D1 | 0.1 (0.22) | 0.0 (0.19)
  EuroQoL Tariffs D252: number analyzed (Participants) | 3 | 6
  EuroQoL Tariffs D252 | -0.4 (0.79) | 0.1 (0.36)
  EuroQoL Tariffs 12M post-D252: number analyzed (Participants) | 65 | 51
  EuroQoL Tariffs 12M post-D252 | 0.0 (0.22) | 0.0 (0.20)
  EuroQoL Tariffs Withdrawal: number analyzed (Participants) | 12 | 15
  EuroQoL Tariffs Withdrawal | -0.2 (0.22) | 0.1 (0.32)

18. Secondary Outcome: PRO - Change From Baseline in HRQL Measures in Participants With FL: The EQ-5D
Description: as for outcome 17
Time Frame: as for outcome 17
Population: Subjects in ITT with FL. ITT population included subjects who were randomized in the study.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 120 | 119
scores on a scale
  EQ5D01-EQ VAS Score C5D1: number analyzed (Participants) | 85 | 76
  EQ5D01-EQ VAS Score C5D1 | 5.5 (19.25) | -6.5 (18.83)
  EQ5D01-EQ VAS Score C11D1: number analyzed (Participants) | 69 | 47
  EQ5D01-EQ VAS Score C11D1 | 12.9 (19.88) | 1.1 (20.87)
  EQ5D01-EQ VAS Score D252: number analyzed (Participants) | 1 | 2
  EQ5D01-EQ VAS Score D252 | 0.00 (NA) — NA = Standard Deviation not available since only 1 participant was analyzed for the assessment | -7.5 (31.82)
  EQ5D01-EQ VAS Score 12M post-D252: number analyzed (Participants) | 46 | 29
  EQ5D01-EQ VAS Score 12M post-D252 | 14.2 (21.47) | 6.7 (20.77)
  EQ5D01-EQ VAS Score Withdrawal: number analyzed (Participants) | 6 | 11
  EQ5D01-EQ VAS Score Withdrawal | -18.5 (13.35) | 5.4 (37.78)
  EuroQoL Tariffs C5D1: number analyzed (Participants) | 84 | 76
  EuroQoL Tariffs C5D1 | 0.0 (0.24) | 0.0 (0.23)
  EuroQoL Tariffs C11D1: number analyzed (Participants) | 70 | 47
  EuroQoL Tariffs C11D1 | 0.1 (0.22) | 0.0 (0.20)
  EuroQoL Tariffs D252: number analyzed (Participants) | 1 | 2
  EuroQoL Tariffs D252 | 0.0 (NA) — NA = Standard Deviation not available since only 1 participant was analyzed for the assessment | 0.4 (0.53)
  EuroQoL Tariffs 12M post-D252: number analyzed (Participants) | 46 | 28
  EuroQoL Tariffs 12M post-D252 | 0.0 (0.22) | 0.0 (0.16)
  EuroQoL Tariffs Withdrawal: number analyzed (Participants) | 6 | 11
  EuroQoL Tariffs Withdrawal | -0.1 (0.16) | 0.1 (0.36)

19. Secondary Outcome: PRO - Change in Health Treatment in HRQL Measures in All Participants: The Health Change Questionnaire (HCQ)
Description: The Health Change Questionnaire,(HCQ) used is a nine item scale that asks the patient to rate change in status since beginning treatment on this study. For HCQ, values from 1 to 9 were assigned to the 9 responses in the HCQ questionnaire, ranging from 1 for 'my health is a great deal better' to 9 for 'my health is a great deal worse' since the beginning of the study. Lower scores represent better conditions
Time Frame: as for outcome 17
Population: ITT: The ITT population included subjects who were randomized in the study.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 173 | 173
scores on a scale
  Change in health treatment C5D1: number analyzed (Participants) | 124 | 118
  Change in health treatment C5D1 | 2.8 (1.81) | 3.8 (2.29)
  Change in health treatment C11D1: number analyzed (Participants) | 105 | 77
  Change in health treatment C11D1 | 2.6 (1.73) | 2.5 (1.74)
  Change in health treatment D252: number analyzed (Participants) | 3 | 6
  Change in health treatment D252 | 5.3 (2.52) | 4.8 (2.56)
  Change in health treatment 12M post D252: number analyzed (Participants) | 66 | 50
  Change in health treatment 12M post D252 | 2.4 (1.95) | 2.6 (1.99)
  Change in health treatment Withdrawal: number analyzed (Participants) | 11 | 15
  Change in health treatment Withdrawal | 5.4 (3.32) | 4.3 (2.63)

20. Secondary Outcome: PRO - Change in Health Treatment in HRQL Measures in Participants With FL: The Health Change Questionnaire (HCQ)
Description: The Health Change Questionnaire, (HCQ) used is a nine item scale that asks the patient to rate change in status since beginning treatment on this study. For HCQ, values from 1 to 9 were assigned to the 9 responses in the HCQ questionnaire, ranging from 1 for 'my health is a great deal better' to 9 for 'my health is a great deal worse' since the beginning of the study. Lower scores represent better conditions
Time Frame: as for outcome 17
Population: Subjects in ITT with FL. ITT population included subjects who were randomized in the study.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 120 | 119
scores on a scale
  Change in health treatment C5D1: number analyzed (Participants) | 86 | 78
  Change in health treatment C5D1 | 2.9 (1.93) | 3.9 (2.25)
  Change in health treatment C11D1: number analyzed (Participants) | 73 | 46
  Change in health treatment C11D1 | 2.7 (1.73) | 2.4 (1.56)
  Change in health treatment D252: number analyzed (Participants) | 1 | 2
  Change in health treatment D252 | 3.0 (NA) — NA: Not enough participants to calculate SD | 4.5 (3.54)
  Change in health treatment 12M post D252: number analyzed (Participants) | 47 | 27
  Change in health treatment 12M post D252 | 2.7 (2.11) | 2.1 (1.54)
  Change in health treatment Withdrawal: number analyzed (Participants) | 5 | 11
  Change in health treatment Withdrawal | 7.2 (1.79) | 4.2 (2.96)

21. Secondary Outcome: Reduction in Tumor Size
Description: Tumor size was measured by the mean change in the sum of the products of the greatest diameter (SPD) of the largest abnormal nodes from baseline to post-baseline by CT Scan.
Time Frame: baseline, post-baseline (up to 55 months)
Population: ITT: The ITT population included subjects who were randomized in the study.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 173 | 173
mm^2 | -33.2 (44.08) | -32.8 (36.83)

22. Secondary Outcome: Summary of Change in Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: This is the number of participants with change in ECOG status. Change is measured categorically by "Improvement, deterioration and No change". Improvement is defined as decrease from baseline by at least one step on the ECOG performance status scale. Deteriorations is defined as increase from baseline by at least one step on the ECOG performance status scale. ECOG status to evaluate daily living: 0: Fully active, able to carry on all pre-disease performance without restriction; 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2: Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3: Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4: Completely disabled; cannot carry on any self care.Totally confined to bed or chai; 5: Dead
Time Frame: as for outcome 17
Population: ITT: The ITT population included subjects who were randomized in the study.
Measure: Number; unit: participants
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 173 | 173
participants
  C5D1: Deteriorated: number analyzed (Participants) | 142 | 134
  C5D1: Deteriorated | 18 | 24
  C5D1: Improved: number analyzed (Participants) | 142 | 134
  C5D1: Improved | 30 | 22
  C5D1: No Change: number analyzed (Participants) | 142 | 134
  C5D1: No Change | 94 | 88
  C11D1: Deteriorated: number analyzed (Participants) | 115 | 90
  C11D1: Deteriorated | 13 | 9
  C11D1: Improved: number analyzed (Participants) | 115 | 90
  C11D1: Improved | 27 | 23
  C11D1: No Change: number analyzed (Participants) | 115 | 90
  C11D1: No Change | 75 | 58
  12M post D252: Deteriorated: number analyzed (Participants) | 70 | 56
  12M post D252: Deteriorated | 9 | 6
  12M post-D252: Improved: number analyzed (Participants) | 70 | 56
  12M post-D252: Improved | 17 | 12
  12M post-D252: No Change: number analyzed (Participants) | 70 | 56
  12M post-D252: No Change | 44 | 38
  Withdrawal: Deteriorated: number analyzed (Participants) | 17 | 21
  Withdrawal: Deteriorated | 7 | 8
  Withdrawal: Improved: number analyzed (Participants) | 17 | 21
  Withdrawal: Improved | 2 | 2
  Withdrawal: No Change: number analyzed (Participants) | 17 | 21
  Withdrawal: No Change | 8 | 11

23. Secondary Outcome: Summary of Number of Participants With Human Anti-Human Antibodies (HAHA)
Description: A summary by responders and non-responders
Time Frame: From randomization up to about 67.5 months
Population: Safety: The Safety population included all subjects who received at least one dose of a study drug. Per protocol, HAHA was only collected for subjects in the Ofa+benda arm.
Measure: Number; unit: Participants
Arm/Group | Ofa + Benda (Arm A)
Number analyzed (Participants) | 151
Participants
  # of participants with post-Ofa HAHA results | 151
  with at least 1 conf. +ve post-Ofa HAHA result | 1
  -ve post-Ofa HAHA results, no Ofa conc. <200 ug/mL | 6
  -ve post-Ofa HAHA, at least 1 Ofa conc<200ug/mL | 144

24. Secondary Outcome: Overall Response Rate (ORR) to Optional Ofatumumab Monotherapy in Subjects Who Progressed During or Following Single-agent Bendamustine
Description: as for outcome 3
Time Frame: From randomization until the 217th PFS event occurred, up to about 67.8 months
Population: ITT: The ITT population included subjects who were randomized in the study.
Measure: Number; unit: Percentage of participants
Groups:
- Optional Ofa: Eligible benda arm participants who were offered optional ofatumumab following disease progression
Arm/Group | Optional Ofa
Number analyzed (Participants) | 30
Percentage of participants | 17

25. Secondary Outcome: Quantitative Assessments of Immunoglobulins A, G and M (IgA, IgG, IgM)
Description: at scheduled visits for actual values as well as for change from baseline
Time Frame: Screening, C1D1, 1M post D252, 6M post D252, 12M post D252 up to 67.5 months; Cycle = 21 days
Population: Safety: The Safety population included all subjects who received at least one dose of a study drug (Ofa+benda arm only).
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Ofa + Benda (Arm A)
Number analyzed (Participants) | 172
g/L
  IgA @ screening (BL): number analyzed (Participants) | 1
  IgA @ screening (BL) | 0.7 (NA) — NA = SD not reached as too few participants
  IgG @ screening: number analyzed (Participants) | 1
  IgG @ screening | 4.7 (NA) — NA = SD not reached as too few participants
  IgM @ screening: number analyzed (Participants) | 1
  IgM @ screening | 0.6 (NA) — NA = SD not reached as too few participants
  IgA @ C1D1: number analyzed (Participants) | 134
  IgA @ C1D1 | 1.3 (0.78)
  IgG @ C1D1: number analyzed (Participants) | 153
  IgG @ C1D1 | 7.7 (3.96)
  IgM @ C1D1: number analyzed (Participants) | 120
  IgM @ C1D1 | 1.4 (4.15)
  IgA @ 1M post-D252: number analyzed (Participants) | 77
  IgA @ 1M post-D252 | 1.1 (0.74)
  IgG @ 1M post-D252: number analyzed (Participants) | 90
  IgG @ 1M post-D252 | 7.1 (2.90)
  IgM @ 1M post-D252: number analyzed (Participants) | 50
  IgM @ 1M post-D252 | 0.6 (0.68)
  IgA @ 6M post D252: number analyzed (Participants) | 65
  IgA @ 6M post D252 | 1.1 (0.59)
  IgG @ 6M post D252: number analyzed (Participants) | 75
  IgG @ 6M post D252 | 7.3 (2.97)
  IgM @ 6M post D252: number analyzed (Participants) | 41
  IgM @ 6M post D252 | 0.7 (0.97)
  IgA @ 12M post D252: number analyzed (Participants) | 53
  IgA @ 12M post D252 | 1.1 (1.2)
  IgG @12M post D252: number analyzed (Participants) | 63
  IgG @12M post D252 | 7.1 (3.31)
  IgM @ 12M post D252: number analyzed (Participants) | 41
  IgM @ 12M post D252 | 0.7 (0.66)

26. Secondary Outcome: Plasma Ofatumumab Concentrations
Description: Concentrations of ofatumumab in plasma listed by actual relative time and summarized by nominal time.
Time Frame: C1D1, C7D1, C12D1, C1D1, C12D1, 12M post-D252, withdrawal up to 12 months follow up
Population: Pharmacokinetic Population: The Pharmacokinetic Population included all subjects who provided at least one evaluable PK concentration
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Ofa + Benda (Arm A)
Number analyzed (Participants) | 171
ug/mL
  C1D1 pre-dose: number analyzed (Participants) | 166
  C1D1 pre-dose | 1.1 (13.97)
  C1D1 End of infusion (EOI): number analyzed (Participants) | 64
  C1D1 End of infusion (EOI) | 262.0 (83.97)
  C1D1 1h post-EOI: number analyzed (Participants) | 61
  C1D1 1h post-EOI | 283.2 (227.11)
  C7D1 pre-dose: number analyzed (Participants) | 128
  C7D1 pre-dose | 153.6 (74.45)
  C7D1 EOI: number analyzed (Participants) | 42
  C7D1 EOI | 402.2 (148.78)
  C7D1 1h post-EOI: number analyzed (Participants) | 39
  C7D1 1h post-EOI | 419.1 (167.44)
  C12D1 pre-dose: number analyzed (Participants) | 101
  C12D1 pre-dose | 143.5 (75.58)
  C12D1 EOI: number analyzed (Participants) | 27
  C12D1 EOI | 392.0 (130.64)
  12M post-D252: number analyzed (Participants) | 43
  12M post-D252 | 0.9 (2.53)
  Withdrawal: number analyzed (Participants) | 13
  Withdrawal | 29.6 (42.58)

27. Secondary Outcome: B-cell Monitoring (CD19+, CD20+)
Description: The percent change of CD5+CD19+ and CD5-CD19+ from baseline was summarized to assess the treatment effect, to monitor the normal B-cell population, and to follow their recovery.
Time Frame: C5D1 (month 5), 1M post-D252, 9M post-D252, up to 67.5 months; Cycle = 21 days
Population: ITT: The ITT population included subjects who were randomized in the study.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 173 | 173
percentage change from baseline
  C5D1: CD45+CD19+: number analyzed (Participants) | 18 | 1
  C5D1: CD45+CD19+ | -94.0 (16.6) | -97.0 (NA) — NA: Not enough participants to calculate SD
  1M post-D252: CD45+CD19+: number analyzed (Participants) | 27 | 0
  1M post-D252: CD45+CD19+ | -82.0 (77.0) |
  9M post-D252: CD45+CD19+: number analyzed (Participants) | 15 | 0
  9M post-D252: CD45+CD19+ | 1421.0 (5721.6) |
  C1D1: CD45+CD20+: number analyzed (Participants) | 17 | 1
  C1D1: CD45+CD20+ | -100.0 (0.0) | -98.0 (NA) — NA: Not enough participants to calculate SD
  1M post-D252: CD45+CD20+: number analyzed (Participants) | 26 | 0
  1M post-D252: CD45+CD20+ | -100.0 (0.0) |
  9M post-D252: CD45+CD20+: number analyzed (Participants) | 15 | 0
  9M post-D252: CD45+CD20+ | 925.0 (3803.1) |

28. Secondary Outcome: Human Anti-chimeric Antibodies (HACA) Over Time
Description: The number of participants with positive and negative baseline HACA results
Time Frame: At Baseline and Cycle 1 day 1
Population: Safety: The Safety population included all subjects who received at least one dose of a study drug
Measure: Number; unit: Participants
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B)
Number analyzed (Participants) | 170 | 142
Participants
  Baseline: Negative | 145 | 119
  Baseline: Positive | 25 | 23
  C1D1: Negative | 145 | 119
  C1D1:Positive | 25 | 23

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) timeframe: Adverse events were collected from first dose of study treatment until end of study treatment plus 60 days, up to maximum duration of 367 days.
Description: AE: Any sign or symptom that occurs during the study treatment plus up to 60 days post treatment
Groups:
- Ofa + Benda (Arm A) + Benda (Arm B) + Optional Ofa: All participants in the Ofa + Benda arm and in the Benda only arm
Arm/Group | Ofa + Benda (Arm A) | Benda (Arm B) | Optional Ofa | Ofa + Benda (Arm A) + Benda (Arm B) + Optional Ofa
All-Cause Mortality (participants affected / at risk) | 66/172 | 71/170 | 15/32 | 137/342
Serious Adverse Events (participants affected / at risk) | 72/172 | 84/170 | 8/32 | 160/342
Other Adverse Events (participants affected / at risk) | 158/172 | 162/170 | 21/32 | 320/342
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofa + Benda (Arm A) (N=172) | Benda (Arm B) (N=170) | Optional Ofa (N=32) | Ofa + Benda (Arm A) + Benda (Arm B) + Optional Ofa (N=342)
Anaemia (Blood and lymphatic system disorders) | 2 | 10 | 0 | 12
Aplastic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 5 | 2 | 15
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 4
Neutropenia (Blood and lymphatic system disorders) | 6 | 8 | 0 | 14
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 6 | 0 | 8
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 2 | 0 | 2
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Optic atrophy (Eye disorders) | 0 | 1 | 0 | 1
Retinal artery occlusion (Eye disorders) | 0 | 1 | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Duodenal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Faecalith (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0 | 3
Asthenia (General disorders) | 1 | 2 | 0 | 3
Death (General disorders) | 3 | 1 | 0 | 4
Disease progression (General disorders) | 0 | 1 | 1 | 2
Fatigue (General disorders) | 1 | 0 | 0 | 1
General physical health deterioration (General disorders) | 1 | 2 | 0 | 3
Malaise (General disorders) | 1 | 2 | 0 | 3
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 2 | 0 | 2
Pyrexia (General disorders) | 7 | 9 | 0 | 16
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 2 | 0 | 2
Type IV hypersensitivity reaction (Immune system disorders) | 0 | 0 | 1 | 1
Abdominal sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Acinetobacter bacteraemia (Infections and infestations) | 1 | 0 | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 1 | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 0 | 1
Candida infection (Infections and infestations) | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 1
Cytomegalovirus chorioretinitis (Infections and infestations) | 1 | 1 | 0 | 2
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 0 | 1
Device related sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Dysentery (Infections and infestations) | 0 | 1 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Febrile infection (Infections and infestations) | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1
Herpes ophthalmic (Infections and infestations) | 0 | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 4 | 0 | 5
Herpes zoster disseminated (Infections and infestations) | 1 | 0 | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1 | 0 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 2
Lung infection (Infections and infestations) | 3 | 2 | 0 | 5
Meningitis (Infections and infestations) | 0 | 1 | 0 | 1
Neutropenic infection (Infections and infestations) | 0 | 1 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 1
Pneumocystis jirovecii infection (Infections and infestations) | 1 | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 2 | 1 | 3
Pneumonia (Infections and infestations) | 10 | 14 | 1 | 25
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 1 | 0 | 1
Postoperative abscess (Infections and infestations) | 1 | 0 | 0 | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 | 1 | 0 | 2
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 3
Sepsis (Infections and infestations) | 1 | 2 | 0 | 3
Septic shock (Infections and infestations) | 1 | 2 | 0 | 3
Sinusitis (Infections and infestations) | 1 | 2 | 0 | 3
Skin infection (Infections and infestations) | 1 | 0 | 0 | 1
Spinal cord infection (Infections and infestations) | 0 | 1 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 1 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 1
Tuberculosis (Infections and infestations) | 1 | 1 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 2
Urosepsis (Infections and infestations) | 1 | 1 | 0 | 2
Varicella (Infections and infestations) | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Cytomegalovirus test positive (Investigations) | 0 | 2 | 0 | 2
Neutrophil count decreased (Investigations) | 2 | 0 | 0 | 2
Oxygen saturation decreased (Investigations) | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 0 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 3
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 2
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0 | 2
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 1
Paraparesis (Nervous system disorders) | 2 | 0 | 0 | 2
Status epilepticus (Nervous system disorders) | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 1
Vascular encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 0 | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 2 | 0 | 3
Urinary tract inflammation (Renal and urinary disorders) | 0 | 1 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 4
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Paraneoplastic pemphigus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Loss of personal independence in daily activities (Social circumstances) | 0 | 1 | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 1
Aortic aneurysm rupture (Vascular disorders) | 1 | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 0 | 1 | 1
Embolism (Vascular disorders) | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 1 | 0 | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ofa + Benda (Arm A) (N=172) | Benda (Arm B) (N=170) | Optional Ofa (N=32) | Ofa + Benda (Arm A) + Benda (Arm B) + Optional Ofa (N=342)
Anaemia (Blood and lymphatic system disorders) | 31 | 46 | 0 | 77
Leukopenia (Blood and lymphatic system disorders) | 25 | 21 | 1 | 46
Lymphopenia (Blood and lymphatic system disorders) | 17 | 17 | 0 | 34
Neutropenia (Blood and lymphatic system disorders) | 66 | 74 | 3 | 141
Thrombocytopenia (Blood and lymphatic system disorders) | 30 | 46 | 1 | 77
Vitreous floaters (Eye disorders) | 1 | 0 | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 9 | 11 | 1 | 20
Constipation (Gastrointestinal disorders) | 29 | 40 | 4 | 72
Diarrhoea (Gastrointestinal disorders) | 35 | 40 | 3 | 75
Dry mouth (Gastrointestinal disorders) | 7 | 9 | 0 | 16
Dyspepsia (Gastrointestinal disorders) | 9 | 7 | 0 | 16
Nausea (Gastrointestinal disorders) | 62 | 93 | 5 | 155
Stomatitis (Gastrointestinal disorders) | 6 | 12 | 1 | 19
Vomiting (Gastrointestinal disorders) | 25 | 40 | 2 | 66
Asthenia (General disorders) | 17 | 27 | 0 | 44
Chills (General disorders) | 9 | 15 | 1 | 25
Fatigue (General disorders) | 41 | 59 | 5 | 101
Influenza like illness (General disorders) | 9 | 4 | 0 | 13
Malaise (General disorders) | 3 | 12 | 0 | 15
Mucosal inflammation (General disorders) | 9 | 14 | 1 | 24
Oedema peripheral (General disorders) | 9 | 14 | 0 | 23
Pyrexia (General disorders) | 33 | 44 | 2 | 78
Bronchitis (Infections and infestations) | 19 | 11 | 0 | 30
Herpes zoster (Infections and infestations) | 9 | 10 | 1 | 20
Nasopharyngitis (Infections and infestations) | 27 | 14 | 1 | 42
Oral herpes (Infections and infestations) | 9 | 10 | 1 | 19
Sinusitis (Infections and infestations) | 10 | 7 | 0 | 17
Upper respiratory tract infection (Infections and infestations) | 12 | 15 | 5 | 29
Urinary tract infection (Infections and infestations) | 11 | 7 | 3 | 21
Infusion related reaction (Injury, poisoning and procedural complications) | 19 | 2 | 4 | 25
Neutrophil count decreased (Investigations) | 13 | 13 | 0 | 26
Platelet count decreased (Investigations) | 12 | 14 | 0 | 26
Weight decreased (Investigations) | 11 | 20 | 0 | 31
White blood cell count decreased (Investigations) | 11 | 9 | 0 | 20
Decreased appetite (Metabolism and nutrition disorders) | 24 | 44 | 2 | 69
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 2 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 8 | 0 | 17
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 15 | 1 | 27
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 12 | 0 | 25
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 5 | 2 | 20
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 2 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 9 | 2 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 8 | 0 | 19
Dizziness (Nervous system disorders) | 14 | 7 | 1 | 22
Dysgeusia (Nervous system disorders) | 9 | 20 | 0 | 29
Headache (Nervous system disorders) | 31 | 21 | 4 | 56
Insomnia (Psychiatric disorders) | 15 | 8 | 3 | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 38 | 27 | 6 | 68
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 21 | 4 | 38
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 3 | 1 | 14
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 4 | 2 | 10
Erythema (Skin and subcutaneous tissue disorders) | 7 | 4 | 2 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 24 | 12 | 4 | 40
Rash (Skin and subcutaneous tissue disorders) | 33 | 15 | 2 | 50
Urticaria (Skin and subcutaneous tissue disorders) | 13 | 1 | 4 | 18
Hypertension (Vascular disorders) | 10 | 6 | 5 | 21
Hypotension (Vascular disorders) | 9 | 6 | 1 | 16
Phlebitis (Vascular disorders) | 6 | 10 | 0 | 16

LIMITATIONS AND CAVEATS:
As the primary endpoint of the study was not met, secondary efficacy endpoints were not fully tested. The data being reported is for information only and not intended to be inferential.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2017-04-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT01077518/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT01077518/SAP_001.pdf